CLINICAL TRIAL: NCT02650310
Title: A New System for Preventing Thermal Stress During Embryo Transfer
Brief Title: New Device to Maintain the Embryo Temperature During Transfer
Acronym: EmbryoTemp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rafael Bernabeu Pérez (Other)
Responsible Party: Sponsor-Investigator, Rafael Bernabeu Pérez, Gynecologist; M D; Ph D, Instituto Bernabeu
Organization: Instituto Bernabeu (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Instituto Bernabeu Group
Record Dates: First submitted 2015-09-28; First posted 2016-01-08 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional transfer (No Intervention): This arm is the control group (conventional embryo transfer protocol) where there is no intervention.
- Thermostable device transfer (Experimental): This arm is the study group: embryo transfer protocol using a new thermostable device.
  Interventions: Device: Thermostable device

INTERVENTIONS:
Device: Thermostable device — Investigators place the catheter with the loaded embryos into a plastic device at 37ºC in order to maintain the temperature
  Arms: Thermostable device transfer

SUMMARY:
The embryo transfer implies transportation from the incubator where they have been at 37 ° C, to the transfer catheter inside a laminar flow hood whose working surface is also maintained at 37 ° C. . From the laboratory to the operating room the embryo is exposed to a temperature drop, and consequently thermal stress occurs, which may compromise its future viability.

The aim of this study is to assess the possible improvement in the clinical results when the embryos are transported in a stable device to avoid the drop in temperature throughout the transfer process.

With the use of this thermosetting device heated to 37 ° C, researchers expect a 15% increase in pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Cryo-transfer cycles: transfer of embryos vitrified in previous cycles receiving donated eggs inseminated with either conjugal or donated sperm from Instituto Bernabeu bank.

Exclusion Criteria:

* Fresh cycles: transfer of fresh embryos (coming from donated or own eggs), and cryo-transfer cycles from vitrified embryos coming from own oocytes.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 352 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-03 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Ongoing Pregnancy rate | Ongoing pregnancy until 28th week of gestation
  Achieving an ongoing pregnancy after embryo transfer

SECONDARY OUTCOMES:
Miscarriage rate | Loss of pregnancy up to 12 weeks of gestation
  To know the embryonic loss rate after implantation
Implantation rate | Embryo implantation after 6-7 weeks of gestation
  To know the embryo implantation rate after the embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Bernabeu, Alicante, Spain